CLINICAL TRIAL: NCT04872907
Title: Prevention of Spontaneous Dental Abscesses in Children With X-linked Hypophosphatemia: a Multicentre Randomized Controlled Trial
Brief Title: Prevention of Spontaneous Dental Abscesses in Children With X-linked Hypophosphatemia : a RCT
Acronym: PRADEX
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: APHP180575
Record Dates: First submitted 2021-03-08; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-03

CONDITIONS: X-linked Hypophosphatemia (XLH)
Keywords: X-linked hypophosphatemia, child, tooth
MeSH Terms: conditions — Familial Hypophosphatemic Rickets | interventions — flowable hybrid composite

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- adhesive system + flowable composite (Experimental): Side of the mouth randomlly assigned to this arm will receive self etch adhesive system and flowable composite combination on temporary molars and self etch adhesive system on anterior temporary teeth at baseline, M6, M12, M18
  Interventions: Device: adhesive system; Drug: flowable composite
- Fluoride varnish (Active Comparator): Side of the mouth randomly assigned to this arm will receive the fluride varnish at baseline, M6, M12, M18 on the temporary teeth
  Interventions: Device: fluoride varnish

INTERVENTIONS:
Device: adhesive system — adhesive system G-BOND. It will be applied to healthy temporary anterior and posterior teeth The adhesive system (on side defined by randomization) will be renew at 6, 12, 18 months, on all three sides due to the physiological wear of the temporary teeth (and therefore the wear of the material).
  Arms: adhesive system + flowable composite
Device: fluoride varnish — The reference drug is a fluoride varnish at 22,600 ppm of the brand Duraphat 50 mg / ml, dental suspension. The varnish is applied to healthy temporary anterior and posterior teeth, on the three sides of the teeth. The reference treatment (on side defined by randomization) will be renew at 6, 12, 18 months, on all three sides due to the physiological wear of the temporary teeth (and therefore the wear of the material).
  Arms: Fluoride varnish
Drug: flowable composite — Composite Essentia HiFlo. It will be applied on healthy temporary molar grooves (on side defined by randomization).
  Complete or partial renewal of the fluid composite in the grooves of the molars in the event of total or partial loss at 6, 12, 18 months
  Arms: adhesive system + flowable composite

SUMMARY:
This study is a prospective, randomized, single-blind, split-mouth, national multicenter trial, comparing the efficacy of a self-etch adhesive system combined (SAM) with a flowable composite to that of a fluoride varnish for the prevention of spontaneous dental abscesses in children with XLH. For each patient, according to randomization, one side of the oral cavity is treated with the experimental treatment (application of the adhesive system to healthy anterior and posterior temporary teeth, and application of the flowable composite to healthy posterior temporary teeth), and the other side with the active comparator (fluoride varnish). The application process for both treatments is similar and will be renewed every 6 months (visits at 6, 12, 18 and 24 months) systematically for the SAM and the varnish, and in case of partial or total loss of the composite.

DETAILED DESCRIPTION:
X-linked hypophosphatemia (XLH) is a vitamin D-resistant familial rickets resulting from a mutation of the PHEX gene. One of the major clinical disorders is dental pulp necrosis, which results in "spontaneous" dental abscesses not related to carious lesions or trauma. These abscesses, which occur in about 67% of children with XLH, can lead to serious complications: loss of teeth, disorders of masticatory, phonetic and aesthetic functions, disorders of occlusion and alveolar-dental development, cervicofacial cellulitis, consequences on the psychological development of the child. this study is the first randomized controlled trial for the prevention of these abscesses.

Primary objective is to evaluate whether a non-invasive adhesive technique, combining the application of a self-etch adhesive system (SAM) to all faces (smooth, proximal and occlusal) of all temporary teeth (anterior and posterior) and a flowable composite applied in the grooves of the posterior temporary teeth, is effective in preventing the development of spontaneous abscesses in children with XLH, compared to the application of a fluoride varnish.

ELIGIBILITY:
Inclusion Criteria:

* X-linked hypophosphatemia diagnosed by the doctor specializing in the disease.
* Patients with at least two healthy contralateral quadrants (right and left) at inclusion defined by the absence of symptomatic or asymptomatic spontaneous abscess, carious lesion and trauma (concussion, subluxation, dislocation, crack, fracture) on all teeth in the quadrant.

Exclusion Criteria:

* Antibiotic treatment within 15 days prior to inclusion
* Patients with a mental disability,
* Patients with cancer, heart disease, sickle cell anemia, pathological bruxism
* Patients with contraindications to study treatments

Ages: 30 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
presence of spontaneous dental abscesses | 24 month after inclusion
  Spontaneous dental abscesses is defined at least one of the following criteria, in the absence of cavities or dental trauma:
  - Clinical criterion: Clinical vestibular, lingual or palatal gingival abscess , or Fistulized abscess, or Fistula, or Head and neck cellulitis .
  - Radiological criteria: Pathological bone radiolucency (periapical or interradicular), visible on a retro-alveolar image.
  The occurrence of at least one spontaneous abscess (binary criterion) will be evaluated for each of the treated sites (4 quadrants per child, corresponding to 2 quadrants on each side of the oral cavity). Only abscesses occurring on a tooth with a history of abscess and free from abscess at inclusion will be considered. Abscesses occurring on a tooth with a carious lesion will not be considered.

SECONDARY OUTCOMES:
Correlation beween the occurrence of spontaneous abscesses and the age at which 1alpha-(OH)D3 was initiated | 24 month after inclusion
infectious complication | 24 month after inclusion
  infectious complication is defined as :sepsis, cavernous sinus thrombophlebitis, mediastinitis, necrotizing fasciits, brain abscess, purulent melting of eye
temporary teeh extracted following a spontaneous abscess on the teeth | 24 month after inclusion

IPD SHARING:
Plan to Share IPD: No